CLINICAL TRIAL: NCT05289219
Title: Effects of Physical Exercise on Sarcopenia After Bariatric Surgery: Protocol of a Randomized Controlled Study
Brief Title: Effects of Physical Exercise on Sarcopenia After Bariatric Surgery
Acronym: EXPOBAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Cláudia Amaro dos Santos, Principal Investigator, University of Évora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21051
Record Dates: First submitted 2022-02-15; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Sarcopenic Obesity; Bariatric Surgery Candidate
Keywords: bariatric surgery; quality of life; metabolic risk factors,; fat-free mass; sarcopenia; exercise
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant
Masking Description: Randomization is performed using a random selection method from the waiting list and the data will be coded and transferred to the database, depending on the intervention group and control group. Data analysis will be done statistically.
  Each participant will be randomly assigned to each group after signing the informed consent and conducting the initial assessments. All laboratory samples and data collected will be identified with identification ID, safeguarding the confidentiality of the collected data.
  At the end of this study, all participants of the control group will be offered the same intervention as the exercise group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The duration of the program is 16-weeks, 3-times a week, for up to 50 minutes per session, starting 1 month after surgery, based on the recommendations of the WHO and the ACSM, because the guidelines for morbidly obese patients undergoing bariatric surgery are not defined. Information on exercises for morbidly obese adults is limited, so the exercise programs will follow the guidelines for adults aged 18 to 65 years healthy, with chronic diseases or disabilities
  Interventions: Behavioral: EXPOBAR
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: EXPOBAR — Each session will start with 5 minutes of warm-up and finalization with 10 minutes of a cool-down, with work of flexibility and proprioception. The maintenance of balance and postural stability may be compromised in obese individuals, depending on the degree of obesity, although the support base provided by the position of the foot is proportional to the structural morphology of each subject. Flexibility is also gradually impaired in obese individuals and of course, these changes may be related to postural changes aggravated by a sedentary lifestyle and biological aging itself alongside all metabolic alterations inherent to the pathology of obesity (Benetti et al., 2016). And the warm-up and the cool-down will be developed as the component of training with the evolution by phases, both in time and in intensity. The first phase will include 20 minutes of interval training, encompassing circuit strength training. Each phase will have an increment of 10 minutes in the central block.
  Arms: Intervention Group

SUMMARY:
The study will include 60 patients awaiting bariatric surgery. They will be randomized into 2 groups, experimental and control. The intervention will take place 1 month after surgery, for a total of 16 weeks. Parameters of body composition, metabolic risk, quality of life, physical activity and sedentary behavior will be determined

DETAILED DESCRIPTION:
Bariatric surgery is the treatment of severe obesity with associated pathologies, with proven evidence in its benefits. Treating overweight allows a better and even reversal of pathologies associated with obesity. In this context, we know that physical exercise is important in the process of weight loss, however, and especially in bariatric surgery, the characteristics of physical activity are not consensual, as well as the effect of programs and physical exercise in this population. Weight loss associated with bariatric surgery is greatly associated with a significant reduction of skeletal muscle and bone mineral mass, which leads us to induce that after bariatric surgery, patients incur an increased risk of sarcopenia. The need for prophylactic programs that prevent sarcopenia in bariatric surgery patients seems to be one of the crucial points for the framing of long-term surgical success of bariatric and metabolic surgery. This randomized clinical trial will aim to study the effects of a 16-week supervised exercise intervention program on the prevention of sarcopenia after bariatric surgery This randomized controlled trial study will include 60 patients of both sexes on the waiting list for bariatric surgery and who have subsequently performed the surgery. They will be randomized into 2 groups, experimental and control. The intervention will take place 1 month after surgery, for a total of 16 weeks. Parameters of body composition, metabolic risk, quality of life, physical activity, and sedentary behavior will be determined.

Assessments will take place in five moments, the surgery, the intervention, the post-intervention, six months after the intervention, twelve months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* As inclusion criteria, patients should be enrolled for bariatric surgery at the hospital
* Aged between 18 years and 60 years
* Contraindication to the practice of exercise
* Agree to participate in the study

Exclusion Criteria:

* Patients with problems in locomotion
* Surgical complications
* Psychiatric diseases and neurological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Body weight | 1 year
  Weight evaluation will be done using a scale
Height | 1 year
  Height evaluation will be done using a stadiometer
Abdominal circumference | 1 year
  Abdominal circumference will be determined by a measuring tape
HDL cholesterol in mg/dl | 1 year
  Blood sample
LDL cholesterol in mg/dl | 1 year
  Blood sample
Triglycerides in mg/dl | 1 year
  Blood sample
Glucose in mg/dl | 1 year
  Blood sample
Insulin in µIU/mL | 1 year
  Blood sample
Glycated hemoglobin in % | 1 year
  Blood sample
Alcohol intake | 1 year
  assessment of daily consumption through clinical data questionnaire
Mean blood pressure | 1 year
  Evaluation with Sphygnomanonetro
Concentration of ghrelin in pg/mg | 1 year
  blood ghrelin and leptin measurement
Concentration of leptin in pg/mg | 1 year
  blood ghrelin and leptin measurement
Lower limbs muscle strength | 1 year
  Lower limbs muscle strength will be evaluated with Biodex
Upper limbs muscle strength | 1 year
  The muscle strength of the upper limbs will be evaluated by manual pressure dynamometry (Handgrip)
Cardiorespiratory fitness | 1 year
  6-minute walk test (TC6)
Cardiorespiratory | 1 year
  Sit-to-stand test for 30 seconds

SECONDARY OUTCOMES:
Life Quality | 1 year
  Questionary "BAROS" as a self-report measure, validated for the Portuguese population specific for bariatric surgery
Salivary amylase | 1 year
  Saliva harvest
physical activity level | 1 year
  Accelerometers measure body movement, providing objective information about the frequency, intensity and duration of physical activity
Glycemia Variation in mg/dl | 1 year
  Evaluation continues through an implantable device for 5 days

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Cláudia Amaro dos Santos, Evora
  - Universidade de Évora, Evora

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baillot A, Mampuya WM, Comeau E, Meziat-Burdin A, Langlois MF. Feasibility and impacts of supervised exercise training in subjects with obesity awaiting bariatric surgery: a pilot study. Obes Surg. 2013 Jul;23(7):882-91. doi: 10.1007/s11695-013-0875-5. PMID 23430477
- [Background] Benetti FA, Bacha IL, Garrido Junior AB, Greve JM. Analyses of balance and flexibility of obese patients undergoing bariatric surgery. Clinics (Sao Paulo). 2016 Feb;71(2):78-81. doi: 10.6061/clinics/2016(02)05. PMID 26934236
- [Background] Broughton DE, Moley KH. Obesity and female infertility: potential mediators of obesity's impact. Fertil Steril. 2017 Apr;107(4):840-847. doi: 10.1016/j.fertnstert.2017.01.017. Epub 2017 Mar 11. PMID 28292619
- [Background] Campbell WW, Kraus WE, Powell KE, Haskell WL, Janz KF, Jakicic JM, Troiano RP, Sprow K, Torres A, Piercy KL, Bartlett DB; 2018 PHYSICAL ACTIVITY GUIDELINES ADVISORY COMMITTEE*. High-Intensity Interval Training for Cardiometabolic Disease Prevention. Med Sci Sports Exerc. 2019 Jun;51(6):1220-1226. doi: 10.1249/MSS.0000000000001934. PMID 31095079
- [Background] Castello V, Simoes RP, Bassi D, Catai AM, Arena R, Borghi-Silva A. Impact of aerobic exercise training on heart rate variability and functional capacity in obese women after gastric bypass surgery. Obes Surg. 2011 Nov;21(11):1739-49. doi: 10.1007/s11695-010-0319-4. PMID 21104041
- [Background] Hanvold SE, Vinknes KJ, Loken EB, Hjartaker A, Klungsoyr O, Birkeland E, Risstad H, Gulseth HL, Refsum H, Aas AM. Does Lifestyle Intervention After Gastric Bypass Surgery Prevent Weight Regain? A Randomized Clinical Trial. Obes Surg. 2019 Nov;29(11):3419-3431. doi: 10.1007/s11695-019-04109-7. PMID 31363961
- [Background] Herring LY, Stevinson C, Carter P, Biddle SJH, Bowrey D, Sutton C, Davies MJ. The effects of supervised exercise training 12-24 months after bariatric surgery on physical function and body composition: a randomised controlled trial. Int J Obes (Lond). 2017 Jun;41(6):909-916. doi: 10.1038/ijo.2017.60. Epub 2017 Mar 6. PMID 28262676
- [Background] Jassil FC, Carnemolla A, Kingett H, Paton B, O'Keeffe AG, Doyle J, Morris S, Lewis N, Kirk A, Pucci A, Chaiyasoot K, Batterham RL. Protocol for a 1-year prospective, longitudinal cohort study of patients undergoing Roux-en-Y gastric bypass and sleeve gastrectomy: the BARI-LIFESTYLE observational study. BMJ Open. 2018 Mar 16;8(3):e020659. doi: 10.1136/bmjopen-2017-020659. PMID 29549212
- [Background] Kalinowski P, Paluszkiewicz R, Wroblewski T, Remiszewski P, Grodzicki M, Bartoszewicz Z, Krawczyk M. Ghrelin, leptin, and glycemic control after sleeve gastrectomy versus Roux-en-Y gastric bypass-results of a randomized clinical trial. Surg Obes Relat Dis. 2017 Feb;13(2):181-188. doi: 10.1016/j.soard.2016.08.025. Epub 2016 Aug 18. PMID 27692906
- [Background] de Oliveira LF, Tisott CG, Silvano DM, Campos CM, do Nascimento RR. GLYCEMIC BEHAVIOR IN 48 HOURS POSTOPERATIVE PERIOD OF PATIENTS WITH TYPE 2 DIABETES MELLITUS AND NON DIABETIC SUBMITTED TO BARIATRIC SURGERY. Arq Bras Cir Dig. 2015;28 Suppl 1(Suppl 1):26-30. doi: 10.1590/S0102-6720201500S100009. PMID 26537269
- [Background] Pekar M, Pekarova A, Buzga M, Holeczy P, Soltes M. The risk of sarcopenia 24 months after bariatric surgery - assessment by dual energy X-ray absorptiometry (DEXA): a prospective study. Wideochir Inne Tech Maloinwazyjne. 2020 Dec;15(4):583-587. doi: 10.5114/wiitm.2020.93463. Epub 2020 Mar 4. PMID 33294073
- [Background] Petta S, Ciminnisi S, Di Marco V, Cabibi D, Camma C, Licata A, Marchesini G, Craxi A. Sarcopenia is associated with severe liver fibrosis in patients with non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2017 Feb;45(4):510-518. doi: 10.1111/apt.13889. Epub 2016 Dec 27. PMID 28028821
- [Background] Soriano-Maldonado A, Martinez-Forte S, Ferrer-Marquez M, Martinez-Rosales E, Hernandez-Martinez A, Carretero-Ruiz A, Villa-Gonzalez E, Barranco-Ruiz Y, Rodriguez-Perez MA, Torrente-Sanchez MJ, Carmona-Rodriguez L, Soriano-Maldonado P, Vargas-Hitos JA, Casimiro-Andujar AJ, Artero EG, Fernandez-Alonso AM. Physical Exercise following bariatric surgery in women with Morbid obesity: Study protocol clinical trial (SPIRIT compliant). Medicine (Baltimore). 2020 Mar;99(12):e19427. doi: 10.1097/MD.0000000000019427. PMID 32195937
- [Background] Villa-Gonzalez E, Barranco-Ruiz Y, Rodriguez-Perez MA, Carretero-Ruiz A, Garcia-Martinez JM, Hernandez-Martinez A, Torrente-Sanchez MJ, Ferrer-Marquez M, Soriano-Maldonado A, Artero EG; EFIBAR Study Group. Supervised exercise following bariatric surgery in morbid obese adults: CERT-based exercise study protocol of the EFIBAR randomised controlled trial. BMC Surg. 2019 Sep 5;19(1):127. doi: 10.1186/s12893-019-0566-9. PMID 31488115
- [Background] Voican CS, Lebrun A, Maitre S, Lainas P, Lamouri K, Njike-Nakseu M, Gaillard M, Tranchart H, Balian A, Dagher I, Perlemuter G, Naveau S. Predictive score of sarcopenia occurrence one year after bariatric surgery in severely obese patients. PLoS One. 2018 May 14;13(5):e0197248. doi: 10.1371/journal.pone.0197248. eCollection 2018. PMID 29758061
- [Derived] Mendes C, Carvalho M, Bravo J, Martins S, Zangao O, Raimundo A. The Impact of an Exercise Program on Health-related Quality of Life (SarQoL) in Patients with Preoperative Sarcopenic Obesity After Bariatric Surgery: A Randomized Controlled Trial. Obes Surg. 2025 Dec;35(12):5000-5012. doi: 10.1007/s11695-025-08326-1. Epub 2025 Nov 26. PMID 41299127
- [Derived] Mendes C, Carvalho M, Cabo CA, Bravo J, Martins S, Raimundo A. Effect of a 16-Week Exercise Program After Bariatric Surgery on Sarcopenia Parameters Based on FNIH, EWGSOP2, and EASO/ESPEN Criteria: the Results of the EXPOBAR Randomized Trial Program. Obes Surg. 2025 Sep;35(9):3553-3568. doi: 10.1007/s11695-025-08142-7. Epub 2025 Aug 13. PMID 40804223